CLINICAL TRIAL: NCT06873321
Title: Incidence of Venous Thromboembolism After Lower Limb Revascularization in Patients Receiving Rivaroxaban 2.5 Mg Bid + Aspirin 100 Mg Versus Single Antiplatelet Treatment - a Randomized Clinical Trial
Brief Title: VTE Incidence After Rivaroxaban + Aspirin or SAPT After Lower-limb Revascularization
Acronym: RESOLUTION
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Science Valley Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CAAE: 77069024.9.0000.8807; CAAE: 77069024.9.0000.8807 (Other: Science Valley)
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Peripheral Arterial Disease; Venous Thormboembolism; Cardiovascular Diseases; Vascular Surgery Patient with PAD / Carotid Stenosis
Keywords: Peripheral Arterial Disease; chronic limb-threatening ischemia; Deep Vein Thrombosis; venous thromboembolism; Factor Xa Inhibitors; rivaroxaban
MeSH Terms: conditions — Peripheral Arterial Disease; Cardiovascular Diseases; Carotid Stenosis; Chronic Limb-Threatening Ischemia; Venous Thrombosis; Venous Thromboembolism | interventions — Rivaroxaban; BID protein, human; Aspirin; Clopidogrel; Endovascular Procedures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Doppler evaluators will be blinded to the study treatment arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study arm (Experimental): Rivaroxaban 2.5 mg bid + aspirin 100 mg
  Interventions: Drug: rivaroxaban 2.5 mg bid + aspirin 100 mg
- comparator (Active Comparator): clopidogrel 75 mg od for 3 months followed by aspirin 100 mg od for endovascular procedures or aspirin for open procedures
  Interventions: Drug: clopidogrel 75 mg od for 3 months followed by aspirin 100 mg od for endovascular procedures or aspirin for open procedures

INTERVENTIONS:
Drug: rivaroxaban 2.5 mg bid + aspirin 100 mg — rivaroxaban 2.5 mg bid + aspirin
  Arms: study arm
Drug: clopidogrel 75 mg od for 3 months followed by aspirin 100 mg od for endovascular procedures or aspirin for open procedures — comparator
  Arms: comparator

SUMMARY:
Venous thromboembolism (VTE) has a high prevalence in patients with multiple comorbidities undergoing complex surgical procedures. Sometimes, extended prophylaxis for VTE with KLMWH or direct oral anticoagulants (DOACs) is necessary. Currently, there is no consensus in the literature regarding the use of DOACs for extended VTE prophylaxis in patients undergoing lower limb revascularization (LLR). Objective: To evaluate the use of DOACs (already approved to reduce MACE and MALE) in VTE prophylaxis in patients undergoing LLR.

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the 30-day VTE incidence in patients submitted to endovascular or open surgery for lower limbs revascularization treated with either rivaroxaban 2.5 mg bid + aspirin 100 mg or single antiplatelet agents (SoC). The main questions it aims to answer are:

Does rivaroxaban 2.5 mg + aspirin reduce the incidence of 30-day VTE?

Researchers will compare rivaroxaban 2.5 mg bid + aspirin 100 mg to a single antiplatelet agent to check comparative VTE incidence.

Participants will:

Take either rivaroxaban 2.5 mg bid + aspirin continuously or single antiplatelet agent (clopidogrel for 3 months followed by aspirin 100 mg for endovascular procedures or aspirin for oper procedures) Visit the clinic once every 2 weeks for checkups and tests, and a mandatory Doppler ultrasound at day 30 Keep a diary of their symptoms

Study Population The study population will consist of patients hospitalized in the vascular surgery ward at the Hospital das Clínicas/Brazilian Hospital Services Company-Federal University of Pernambuco (HC/EBSERH-UFPE) who undergo arterial revascularization surgery of the lower limbs (LL) via angioplasty (ATP) or bypass surgery.

The study will determine the sample size by the criteria established by Resolution 466/12 of the National Health Council. The estimated sample size is 200 research participants, with 100 in the study group and 100 in the control group. If the degree of dispersion is high, the number of research participants may be adjusted.

Study Design A single-center randomized clinical trial. Randomization will be performed using the REDCap platform. Due to the nature of the procedure, blinding will not be possible.

Considering an acceptable margin of error (5%), a confidence level of 95%, and a prevalence of 50% for venous diseases, with a heterogeneity level of 50%.

Selection of Research Participants The selection of research participants will follow specific inclusion and exclusion criteria. After selection, participants will be randomly assigned to the Study Group (SG) or the Control Group (CG).

CG (Control Group): Will receive standard treatment as described in the literature: Aspirin (ASA) 100 mg once daily for patients undergoing lower limb bypass revascularization, and ASA 100 mg once daily combined with Clopidogrel 75 mg once daily for patients undergoing lower limb angioplasty.

SG (Study Group): Will receive ASA 100 mg once daily plus Rivaroxaban 2.5 mg twice daily for patients undergoing bypass or angioplasty revascularization.

A total of 100 patients will be included in the study, equally divided between the control and study groups. Randomization will be performed via the REDCap platform.

ELIGIBILITY:
Inclusion Criteria:

1. Be adults of any age and gender.
2. Have critical limb ischemia with a proposed revascularization treatment (either via ATP or bypass surgery) at the Vascular Surgery Service of HC/EBSERH - UFPE.
3. Sign the informed consent form (ICF) (Appendix 2).

Exclusion Criteria:

1. Experience a symptomatic VTE event during hospitalization, as they will require full anticoagulation rather than prophylactic anticoagulation.
2. Have any contraindications to Rivaroxaban.
3. Do not return for the 30-day postoperative follow-up visit.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-24 (Actual); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
primary efficacy outcome | 30 days
  Incidence of symptomatic + asymptomatic deep vein thrombosis (DVT) or pulmonary embolism (PE) 30 days post-hospital discharge.
primary safety outcome | 30 days
  Combination of clinically relevant non-major bleeding + major bleeding defined by the ISTH criteria

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Ramacciotti, MD, Ph.D., Study Director — Science Valley
Locations (1):
- Hospital das Clínicas, Federal University of Pernambuco, Pernambuco, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Anonymized participant data can be made available upon requests directed to the corresponding author. Proposals will be reviewed based on scientific merit. After a proposal is approved, data can be shared through a secure online platform after signing a data access agreement.

REFERENCES:
- [Background] Bonaca MP, Bauersachs RM, Anand SS, Debus ES, Nehler MR, Patel MR, Fanelli F, Capell WH, Diao L, Jaeger N, Hess CN, Pap AF, Kittelson JM, Gudz I, Matyas L, Krievins DK, Diaz R, Brodmann M, Muehlhofer E, Haskell LP, Berkowitz SD, Hiatt WR. Rivaroxaban in Peripheral Artery Disease after Revascularization. N Engl J Med. 2020 May 21;382(21):1994-2004. doi: 10.1056/NEJMoa2000052. Epub 2020 Mar 28. PMID 32222135
- [Background] Eikelboom JW, Connolly SJ, Bosch J, Dagenais GR, Hart RG, Shestakovska O, Diaz R, Alings M, Lonn EM, Anand SS, Widimsky P, Hori M, Avezum A, Piegas LS, Branch KRH, Probstfield J, Bhatt DL, Zhu J, Liang Y, Maggioni AP, Lopez-Jaramillo P, O'Donnell M, Kakkar AK, Fox KAA, Parkhomenko AN, Ertl G, Störk S, Keltai M, Ryden L, Pogosova N, Dans AL, Lanas F, Commerford PJ, Torp-Pedersen C, Guzik TJ, Verhamme PB, Vinereanu D, Kim JH, Tonkin AM, Lewis BS, Felix C, Yusoff K, Steg PG, Metsarinne KP, Cook Bruns N, Misselwitz F, Chen E, Leong D, Yusuf S; COMPASS Investigators. Rivaroxaban with or without Aspirin in Stable Cardiovascular Disease. N Engl J Med. 2017 Oct 5;377(14):1319-1330. doi: 10.1056/NEJMoa1709118. Epub 2017 Aug 27. PMID: 28844192. Copy
- [Background] Gould MK, Garcia DA, Wren SM, Karanicolas PJ, Arcelus JI, Heit JA, Samama CM. Prevention of VTE in nonorthopedic surgical patients: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e227S-e277S. doi: 10.1378/chest.11-2297. PMID 22315263
- [Background] Haykal T, Zayed Y, Kerbage J, Deliwala S, Long CA, Ortel TL. Meta-analysis and systematic review of randomized controlled trials assessing the role of thromboprophylaxis after vascular surgery. J Vasc Surg Venous Lymphat Disord. 2022 May;10(3):767-777.e3. doi: 10.1016/j.jvsv.2021.08.019. Epub 2021 Sep 8. PMID 34508872
- [Background] Dagher NN, Modrall JG. Pharmacotherapy before and after revascularization: anticoagulation, antiplatelet agents, and statins. Semin Vasc Surg. 2007 Mar;20(1):10-4. doi: 10.1053/j.semvascsurg.2007.02.006. PMID 17386359
- [Background] Chindamo MC, Marques MA. Bleeding risk assessment for venous thromboembolism prophylaxis. J Vasc Bras. 2021 Apr 28;20:e20200109. doi: 10.1590/1677-5449.200109. PMID 34093680
- [Derived] de Oliveira Buril G, Portugal MF, Neves S, da Silva VS, Sad EF, Caffaro RA, Volpiani GG, Bernardi WH, Leal IZ, Pimentel TF, Simoni GH, Lins EM, Ramacciotti E. Venous Thromboembolism in Patients Receiving Rivaroxaban Plus Aspirin or Standard Treatment after Lower Limb Revascularization-Rationale and Design of the RESOLUTION Trial. Ann Vasc Surg. 2025 Nov 11;124:22-27. doi: 10.1016/j.avsg.2025.10.041. Online ahead of print. PMID 41232756